CLINICAL TRIAL: NCT01747629
Title: A 12-week Comparison of the Efficacy and Safety and Steady-State Pharmacokinetics of Albuterol Spiromax® Versus Placebo in Subjects 12 Years and Older With Persistent Asthma
Brief Title: Efficacy of Inhaled Albuterol Spiromax® in Subjects With Persistent Asthma With Steady State Pharmacokinetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABS-AS-304
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-05

CONDITIONS: Asthma
Keywords: Asthma; dry powder inhaler; short-acting beta2-agonist; SABA; bronchoconstriction; bronchodilation; bronchodilator; metered dose inhaler; Albuterol Spiromax®
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo MDPI (Placebo Comparator): Placebo multi-dose dry powder inhaler (MDPI) administered as 2 inhalations four times a day for 12 weeks.
  Interventions: Drug: Placebo MDPI
- Albuterol MDPI (Experimental): Albuterol multi-dose dry powder inhaler (MDPI) at a dose of 720 micrograms per day administered as 2 inhalations of 90 mcg /inhalation four times a day for 12 weeks.
  Interventions: Drug: Albuterol MDPI

INTERVENTIONS:
Drug: Placebo MDPI — Placebo MDPI administered as 2 inhalations 4 times a day (QID) (at approximately 7:00 AM, 12 noon, 5:00 PM, and bedtime) for 12 weeks.
  Other Names: Placebo Spiromax®
  Arms: Placebo MDPI
Drug: Albuterol MDPI — Albuterol MDPI administered as 2 inhalations 4 times a day (QID) (at approximately 7:00 AM, 12 noon, 5:00 PM, and bedtime) for 12 weeks.
  Other Names: ProAir® RespiClick, Albuterol Spiromax®
  Arms: Albuterol MDPI

SUMMARY:
The primary objective of this study is to evaluate the efficacy of Albuterol Spiromax® versus placebo in subjects with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent
* At least 12 years of age at screening
* General good health
* Persistent asthma for ≥3 months, with an FEV1 50-80% predicted and ≥15% reversibility
* Taking inhaled corticosteroids at a stable dose (≤ equivalent of 500mcg of fluticasone propionate/day) for at least 4 weeks prior to the Screening Visit.
* Ability to perform spirometry in an acceptable manner as per protocol guidelines
* Other inclusion criteria apply

Exclusion Criteria:

* A known hypersensitivity to albuterol or any of the excipients in the formulations.
* History of a respiratory infection or disorder that has not resolved within 1 week preceding the Screening Visit (SV).
* History of life-threatening asthma that is defined for this protocol as an asthma episode that required intubation.
* Any asthma exacerbation requiring oral corticosteroids within 3 months of the SV. A subject must not have had any hospitalization for asthma within 6 months prior to the SV.
* Hospitalization due to asthma exacerbation 2 or more times in the past year
* Initiation of immunotherapy or dose escalation during the study period
* Other exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Leader, Study Director — Teva Respiratory R&D
Locations (35):
- United States (35):
  - Teva Investigational Site 10225, Costa Mesa, California
  - Teva Investigational Site 10250, Encinitas, California
  - Teva Investigational Site 10230, Huntington Beach, California
  - Teva Investigational Site 10255, Palmdale, California
  - Teva Investigational Site 10231, Rancho Mirage, California
  - Teva Investigational Site 10252, Riverside, California
  - Teva Investigational Site 10242, Rolling Hills Estates, California
  - Teva Investigational Site 10238, San Diego, California
  - Teva Investigational Site 10243, San Jose, California
  - Teva Investigational Site 10247, Miami Lakes, Florida
  - Teva Investigational Site 10239, Tallahassee, Florida
  - Teva Investigational Site 10234, Tampa, Florida
  - Teva Investigational Site 10253, Bangor, Maine
  - Teva Investigational Site 10257, Baltimore, Maryland
  - Teva Investigational Site 10254, White Marsh, Maryland
  - Teva Investigational Site 10235, Fall River, Massachusetts
  - Teva Investigational Site 10236, North Dartmouth, Massachusetts
  - Teva Investigational Site 10226, Minneapolis, Minnesota
  - Teva Investigational Site 10233, Minneapolis, Minnesota
  - Teva Investigational Site 10241, St Louis, Missouri
  - Teva Investigational Site 10229, Bellevue, Nebraska
  - Teva Investigational Site 10227, Rochester, New York
  - Teva Investigational Site 10244, Charlotte, North Carolina
  - Teva Investigational Site 10248, Cincinnati, Ohio
  - Teva Investigational Site 10249, Oklahoma City, Oklahoma
  - Teva Investigational Site 10232, Eugene, Oregon
  - Teva Investigational Site 10259, Medford, Oregon
  - Teva Investigational Site 10237, Portland, Oregon
  - Teva Investigational Site 10240, Bethlehem, Pennsylvania
  - Teva Investigational Site 10246, Pittsburgh, Pennsylvania
  - Teva Investigational Site 10256, Pittsburgh, Pennsylvania
  - Teva Investigational Site 10251, Rock Hill, South Carolina
  - Teva Investigational Site 10228, Spartanburg, South Carolina
  - Teva Investigational Site 10258, San Antonio, Texas
  - Teva Investigational Site 10245, Seattle, Washington

REFERENCES:
- [Derived] Raphael G, Taveras H, Iverson H, O'Brien C, Miller D. Twelve- and 52-week safety of albuterol multidose dry powder inhaler in patients with persistent asthma. J Asthma. 2016;53(2):187-93. doi: 10.3109/02770903.2015.1070862. Epub 2015 Sep 15. PMID 26369589

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 361 patients screened, 158 were excluded on the basis of inclusion criteria, 5 on the basis of exclusion criteria, 13 withdrew consent, 1 patient was noncompliant, 2 patients were lost to follow-up before the baseline visit, 7 patients had other reasons, and 15 failed to meet the randomization criteria at the end of the run-in period.
Period: Overall Study
Arm/Group | Placebo MDPI | Albuterol MDPI
Started | 85 | 75
Treated | 84 (Safety set and full analysis set) | 75 (Safety set and full analysis set)
Completed | 77 | 69
Not Completed | 8 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Noncompliance | 1 | 1
Not completed — Inclusion criteria not met | 1 | 0
Not completed — Not treated | 1 | 0
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: Randomized analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo MDPI | Albuterol MDPI | Total
Number analyzed (Participants) | 85 | 75 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (15.94) | 40.0 (18.06) | 38.2 (16.99)
Age, Customized [Number; unit: participants]
  12-17 years | 17 | 14 | 31
  18-64 years | 67 | 58 | 125
  65+ years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 36 | 81
  Male | 40 | 39 | 79
Race/Ethnicity, Customized [Number; unit: participants]
  White | 66 | 59 | 125
  Black | 17 | 11 | 28
  Asian | 1 | 0 | 1
  American Indian or Alaskan Native | 0 | 1 | 1
  Pacific Islander | 0 | 1 | 1
  Other | 1 | 3 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 77 | 69 | 146
Weight [Mean (Standard Deviation); unit: kg] | 79.8 (22.76) | 79.6 (20.75) | 79.7 (21.77)
Height [Mean (Standard Deviation); unit: cm] | 167.8 (9.23) | 169.8 (10.93) | 168.7 (10.08)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.1 (6.48) | 27.4 (5.90) | 27.7 (6.21)

OUTCOME MEASURES:

1. Primary Outcome: Baseline-adjusted Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC 0-6) Over the 12-week Treatment Period
Description: FEV1 AUC 0-6 is the area under the effect-time curve from time 0 (pre-dose) up to 6 hours post-dose. It represents the weighted average (by the trapezoidal rule) over six hours of the FEV1 AUC 0-6 measures adjusted for the baseline measure (i.e., change from baseline at each timepoint) recorded on days 1, 8 and 85 of the treatment period. The baseline for each study day was the average of the 2 pre-dose FEV1 measurements on that study day.
  FEV1 was measured using spirometry. Spirometry assessments were obtained predose at -30 ± 5, and - 5 minutes, then post dose at 5 ± 2, 15 ± 5, 30 ± 5, 45 ± 5 minutes, and at 1hr ± 5 min, 2hr ± 5 min, 3hr ± 5 min, 4hr ± 5 min, 5hr ± 5 min, and 6hr ± 5 min.
Time Frame: Day 1, Day 8 and Day 85
Population: Full analysis set included all participants in the intent-to-treat population who received at least 1 dose of study medication and had at least 1 post-baseline assessment.
Measure: Mean (Standard Error); unit: L*hr
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 84 | 75
L*hr | 0.38 (0.114) | 1.30 (0.120)
Statistical Analysis 1: Comparison: Placebo MDPI vs Albuterol MDPI; Test type: Superiority or Other; p < 0.0001, mixed-model repeated-measures (MMRM) — Significance at the 0.05 level; Fixed effects- pooled center, treatment group, study day, and study day by drug interaction, with baseline measured at each study day as covariate; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [0.59 to 1.24], Standard Error of Mean 0.163

2. Secondary Outcome: Baseline-adjusted Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC 0-6) on Day 1
Description: FEV1 AUC 0-6 is the area under the effect-time curve from time 0 (pre-dose) up to 6 hours post-dose. It represents the weighted average over six hours of the FEV1 AUC 0-6 measures adjusted for the baseline measure. The baseline was the average of the 2 pre-dose FEV1 measurements on that study day.
  FEV1 was measured using spirometry. Spirometry assessments were obtained predose at -30 ± 5, and - 5 minutes, then post dose at 5 ± 2, 15 ± 5, 30 ± 5, 45 ± 5 minutes, and at 1hr ± 5 min, 2hr ± 5 min, 3hr ± 5 min, 4hr ± 5 min, 5hr ± 5 min, and 6hr ± 5 min.
Time Frame: Day 1
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: L*hr
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 84 | 75
L*hr | 0.58 [0.24 to 0.92] | 1.63 [1.27 to 1.99]
Statistical Analysis 1: Comparison: Placebo MDPI vs Albuterol MDPI; Test type: Superiority or Other; p < 0.0001, mixed model repeated measures (MMRM) — To adjust for multiplicity, so that the overall alpha level for all tests was controlled at the 0.05 level, tests were done sequentially [day 1, then day 8, then day 85] and terminated if individual results were not significant at the 0.05 level; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.05, 95% CI 2-sided [0.56 to 1.55], Standard Error of Mean 0.249

3. Secondary Outcome: Baseline-adjusted Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC 0-6) on Day 8
Description: as for outcome 2
Time Frame: Day 8
Population: Full analysis set of participants with data at the time point
Measure: Mean (95% Confidence Interval); unit: L*hr
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 83 | 74
L*hr | 0.37 [0.08 to 0.66] | 1.15 [0.84 to 1.45]
Statistical Analysis 1: Comparison: Placebo MDPI vs Albuterol MDPI; Test type: Superiority or Other; p = 0.0004, mixed model repeated measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [0.35 to 1.19], Standard Error of Mean 0.212

4. Secondary Outcome: Baseline-adjusted Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC 0-6) on Day 85
Description: as for outcome 2
Time Frame: Day 85
Population: Full analysis set of participants with data at the time point
Measure: Mean (95% Confidence Interval); unit: L*hr
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 78 | 69
L*hr | 0.20 [-0.05 to 0.44] | 1.12 [0.86 to 1.38]
Statistical Analysis 1: Comparison: Placebo MDPI vs Albuterol MDPI; Test type: Superiority or Other; p < 0.0001, mixed model repeated measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.93, 95% CI 2-sided [0.57 to 1.28], Standard Error of Mean 0.180

5. Secondary Outcome: Participants With Adverse Events
Description: Adverse events (AEs) summarized in this table are those that began or worsened after treatment with study drug (treatment-emergent AEs). An adverse event was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to Day 93
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 84 | 75
participants
  Any adverse event | 36 | 22
  Severe adverse event | 3 | 1
  Treatment-related adverse event | 2 | 1
  Deaths | 0 | 0
  Other serious adverse event | 0 | 2
  Withdrawn from study due to adverse event | 1 | 2

6. Secondary Outcome: Physical Examination Findings Shifts From Baseline to Endpoint by Treatment Group
Description: Physical exam was recorded as normal or abnormal based on physician assessment. Format for results is: Test Baseline/Endpoint. HEENT = head, eyes, ears, nose, throat.
Time Frame: Day 1 (Baseline), Day 85
Population: Safety population. Only participants with both baseline and endpoint physical examination findings are summarized.
Measure: Number; unit: participants
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 84 | 75
participants
  General appearance Normal/Normal | 81 | 72
  General appearance Normal/Abnormal | 0 | 1
  General appearance Abnormal/Normal | 0 | 0
  General appearance Abnormal/Abnormal | 2 | 1
  HEENT Normal/Normal | 59 | 52
  HEENT Normal/Abnormal | 1 | 2
  HEENT Abnormal/Normal | 7 | 5
  HEENT Abnormal/Abnormal | 16 | 15
  Chest and Lungs Normal/Normal | 76 | 64
  Chest and Lungs Normal/Abnormal | 2 | 3
  Chest and Lungs Abnormal/Normal | 3 | 7
  Chest and Lungs Abnormal/Abnormal | 2 | 0
  Heart Normal/Normal | 82 | 70
  Heart Normal/Abnormal | 0 | 1
  Heart Abnormal/Normal | 0 | 0
  Heart Abnormal/Abnormal | 1 | 3
  Abdomen Normal/Normal | 82 | 71
  Abdomen Normal/Abnormal | 0 | 1
  Abdomen Abnormal/Normal | 0 | 0
  Abdomen Abnormal/Abnormal | 1 | 2
  Musculoskeletal Normal/Normal | 81 | 72
  Musculoskeletal Normal/Abnormal | 1 | 1
  Musculoskeletal Abnormal/Normal | 0 | 0
  Musculoskeletal Abnormal/Abnormal | 1 | 1
  Skin Normal/Normal | 69 | 63
  Skin Normal/Abnormal | 5 | 1
  Skin Abnormal/Normal | 2 | 4
  Skin Abnormal/Abnormal | 7 | 6
  Lymph nodes Normal/Normal | 83 | 74
  Lymph nodes Normal/Abnormal | 0 | 0
  Lymph nodes Abnormal/Normal | 0 | 0
  Lymph nodes Abnormal/Abnormal | 0 | 0
  Neurological Normal/Normal | 83 | 74
  Neurological Normal/Abnormal | 0 | 0
  Neurological Abnormal/Normal | 0 | 0
  Neurological Abnormal/Abnormal | 0 | 0

7. Secondary Outcome: Participants With Clinically Significant Vital Sign Assessments
Description: For both standard and serial vital signs, participants were seated for at least 5 minutes before vital signs were assessed. Heart rate was obtained prior to the blood pressure measurement. Serial heart rate and blood pressure were conducted in the sitting position prior to the spirometry assessment; baseline measures were taken pre-dose at -30 ± 5 and -5 minutes on Day 1. Day 85 serial vital sign measures were taken in the sitting position prior to spirometry assessments pre-dose at -30 ± 5 and -5 minutes, then post-dose at 30 (±5) minutes, 1hr (± 10 min), 2hr (± 10 min), 3hr (± 10 min), 4hr (± 10 min), 5hr (± 10 min) and 6 hr (± 10 min).
  Serial heart rate and blood pressure measurements that were elevated to the following criteria were considered clinically significant:
  Systolic blood pressure: > 160 beats/minute Diastolic blood pressure: >100 beats/minute Heart rate: >120 beats/minute
Time Frame: Days 8 and 85
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 84 | 75
participants
  Systolic blood pressure - high | 2 | 3
  Diastolic blood pressure - high | 2 | 2
  Heart rate - high | 0 | 0

8. Secondary Outcome: Maximum Observed Plasma Drug Concentration (Cmax) for Albuterol on Days 1 and 8
Description: Pharmacokinetic parameters of albuterol were determined on Day 1 after the first dose administration and at steady-state on Day 8. Day 1 serial (10-hr) blood samples for pharmacokinetics pre-dose (within 30 minutes prior to dosing), and post-dose at the following times: 15 (±5) min, 30 (±5) min, and 1, 2, 3, 4, 5, 6, 8 and 10 hours (±10 minutes). Day 8 serial (6-hr) blood samples for pharmacokinetics pre-dose (within 30 min prior to dosing), and post-dose at the following times: 15 (±5) min, 30 (±5) min, and 1, 2, 3, 4, 5 and 6 hr (±10 min).
Time Frame: Days 1 and 8
Population: Pharmacokinetic analysis set representing a subset of participants from the Albuterol MDPI treatment arm.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 0 | 16
pg/mL
  Day 1 |  | 347.2 (146.6)
  Day 8 |  | 499.1 (154.3)

9. Secondary Outcome: Time to Observed Peak Plasma Concentration (Tmax) for Albuterol on Days 1 and 8
Description: as for outcome 8
Time Frame: Days 1 and 8
Population: Pharmacokinetic analysis set representing a subset of participants from the Albuterol MDPI treatment arm.
Measure: Median (Full Range); unit: hour
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 0 | 16
hour
  Day 1 |  | 0.48 [0.18 to 4.95]
  Day 8 |  | 0.44 [0.25 to 2.02]

10. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 (Pre-dose) up to 6 Hours Post-dose (AUC0-6) for Albuterol on Days 1 and 8
Description: Pharmacokinetic parameters of albuterol were determined on Day 1 after the first dose administration and at steady-state on Day 8. Day 1 serial (10-hr) blood samples for pharmacokinetics pre-dose (within 30 minutes prior to dosing), and post-dose at the following times: 15 (±5) min, 30 (±5) min, and 1, 2, 3, 4, 5, 6, 8 and 10 hours (±10 minutes). Day 8 serial (6-hr) blood samples for pharmacokinetics pre-dose (within 30 min prior to dosing), and post-dose at the following times: 15 (±5) min, 30 (±5) min, and 1, 2, 3, 4, 5 and 6 hr (±10 min).
  AUC0-6 on Day 8 is not from pre-dose but at steady state.
Time Frame: Days 1 and 8
Population: Pharmacokinetic analysis set representing a subset of participants from the Albuterol MDPI treatment arm.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 0 | 16
pg*hr/mL
  Day 1 |  | 1325 (646)
  Day 8 |  | 2163 (825)

11. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 (Pre-dose) to Last Time of Quantifiable Concentration (AUC0-t) for Albuterol on Days 1 and 8
Description: Pharmacokinetic parameters of albuterol were determined on Day 1 after the first dose administration and at steady-state on Day 8. Day 1 serial (10-hr) blood samples for pharmacokinetics pre-dose (within 30 minutes prior to dosing), and post-dose at the following times: 15 (±5) min, 30 (±5) min, and 1, 2, 3, 4, 5, 6, 8 and 10 hours (±10 minutes). Day 8 serial (6-hr) blood samples for pharmacokinetics pre-dose (within 30 min prior to dosing), and post-dose at the following times: 15 (±5) min, 30 (±5) min, and 1, 2, 3, 4, 5 and 6 hr (±10 min).
  AUC0-t on Day 8 is not from pre-dose but at steady state.
Time Frame: Days 1 and 8
Population: Pharmacokinetic analysis set representing a subset of participants from the Albuterol MDPI treatment arm.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 0 | 16
pg*hr/mL
  Day 1 |  | 1747 (785)
  Day 8 |  | 2165 (839)

12. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 (Pre-dose) to Infinity Post-dose(AUC0-inf) for Albuterol on Day 1
Description: as for outcome 8
Time Frame: Day 1
Population: Pharmacokinetic analysis set representing a subset of participants from the Albuterol MDPI treatment arm.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 0 | 16
pg*hr/mL |  | 2278 (869)

13. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 (Pre-dose) to 24 Hours Post-dose(AUC0-24) for Albuterol on Day 8
Description: as for outcome 8
Time Frame: Day 8
Population: Pharmacokinetic analysis set representing a subset of participants from the Albuterol MDPI treatment arm.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 0 | 16
pg*hr/mL |  | 3605 (1189)

14. Secondary Outcome: Terminal Plasma Half-life (t1/2) for Albuterol on Days 1 and 8
Description: as for outcome 8
Time Frame: Days 1 and 8
Population: Pharmacokinetic analysis set representing a subset of participants from the Albuterol MDPI treatment arm.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 0 | 16
hour
  Day 1 |  | 4.7 (1.3)
  Day 8 |  | 5.7 (1.4)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 93
Arm/Group | Albuterol MDPI | Placebo MDPI
Serious Adverse Events (participants affected / at risk) | 2/75 | 0/84
Other Adverse Events (participants affected / at risk) | 9/75 | 10/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albuterol MDPI (N=75) | Placebo MDPI (N=84)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albuterol MDPI (N=75) | Placebo MDPI (N=84)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 2 (2)
Headache (Nervous system disorders) | 1 (2) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.